CLINICAL TRIAL: NCT07385911
Title: Olfactory Outcomes of Cautery Vs Scalpel in Endoscopic Endonasal Skull Base Surgery- A Prospective Randomised Controlled Study.
Brief Title: A Clinical Trial to Study the Effects on the Olfaction Capacity of an Individual Undergoing Skull Base Surgeries Using Cautery vs Scalpel .
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Jodhpur (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIIMS/IEC/2025/5462
Record Dates: First submitted 2025-12-18; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Olfaction
MeSH Terms: conditions — Anosmia | interventions — Laser Therapy; Cautery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): During endoscopic endonasal skull base surgery,scalpel will be used to elevate the nasoseptal flap.
  Interventions: Procedure: Scalpel
- Group B (Active Comparator): During endoscopic endonasal skull base surgery,cautery will be used to elevate the nasoseptal flap.
  Interventions: Procedure: Cautery

INTERVENTIONS:
Procedure: Scalpel — During endoscopic endonasal skull base surgery,scalpel will be used to elevate the nasoseptal flap.
  Arms: Group A
Procedure: Cautery — During endoscopic endonasal skull base surgery,cautery will be used to elevate the nasoseptal flap.
  Arms: Group B

SUMMARY:
Olfaction is a prominent entity that determines a person's quality of life. During human evolution, olfaction has played an essential role in determining safe food, assessing threats, and developing social relationships. Endoscopic endonasal surgeries are widely used today for the removal of brain tumors involving the pituitary and skull base. The minimal invasiveness, rapid recovery, better visualization, and lower occurrence of complication make endonasal endoscopic surgery an ideal approach for tumors involving the pituitary and midline skull base. However, the olfactory epithelium is at risk of injury during endoscopic skull base surgeries due to the orientation of the olfactory epithelium fibers.It has been found that the olfactory neuroepithelium extends from the cribriform plate superiorly to the septum for the superior-most 1 to 2 cm medially and onto the upper half of the superior turbinates laterally.It also extends from the face of the sphenoid posteriorly to the attachment of the middle turbinate anteriorly.This makes the olfactory fibers susceptible to injury during endonasal surgery that requires superior or upper limb septal incisions, such as the pedicled nasoseptal flap (the Hadad-Bassagasteguy flap) and modified nasoseptal rescue flap.It has been debated whether using a scalpel instead of cautery could have a differential effect on the olfaction of an individual, as some surgeons believe that the heat generated by a cautery injures the nearby olfactory mucosa.This study aims at determining the method which is better at preserving the olfactory capacity of an individual undergoing endoscopic endonasal skull base surgery.

ELIGIBILITY:
Inclusion Criteria:

-Patients undergoing endoscopic endonasal skull base surgeries that require the raising of a nasoseptal flap

Exclusion Criteria:

* Patients with preoperative anosmia due to any cause.
* Patients with a previous history of sino-nasal, pituitary, or skull base surgery.
* Patients with a medical history of neurodegenerative diseases (for example, Alzheimer's disease or Parkinson's disease), chronic rhinosinusitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Combined Olfactory Score (I-smell test) | Preoperatively,Immediate postoperatively,3-6 months postoperatively
  Threshold odour identification score and specific odour identification score will be added to form a Combined Olfactory Score.
Visual Analogue Scale (VAS) | Preoperatively,Immediately postoperatively,3-6 months postoperatively
  Visual analogue scale scoring from 0-10 to measure olfaction. (with higher score indicating better olfaction capacity)

SECONDARY OUTCOMES:
22-item Sino Nasal Outcome Test (SNOT-22) questionnaire | Preoperatively,Immediate postoperatively,3-6 months postoperatively
  It covers a range of sinonasal symptoms and their impact on social and emotional well-being

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute Of Medical Sciences, Jodhpur, Rajasthan, India

REFERENCES:
- [Result] Kim SW, Park KB, Khalmuratova R, Lee HK, Jeon SY, Kim DW. Clinical and histologic studies of olfactory outcomes after nasoseptal flap harvesting. Laryngoscope. 2013 Jul;123(7):1602-6. doi: 10.1002/lary.24107. Epub 2013 Mar 21. PMID 23798331
- [Result] Puccinelli CL, Yin LX, O'Brien EK, Van Gompel JJ, Choby GW, Van Abel KM, Janus JR, Stokken JK. Long-term olfaction outcomes in transnasal endoscopic skull-base surgery: a prospective cohort study comparing electrocautery and cold knife upper septal limb incision techniques. Int Forum Allergy Rhinol. 2019 May;9(5):493-500. doi: 10.1002/alr.22291. Epub 2019 Jan 18. PMID 30657649
- [Result] Hong SD, Nam DH, Park J, Kim HY, Chung SK, Dhong HJ. Olfactory outcomes after endoscopic pituitary surgery with nasoseptal "rescue" flaps: electrocautery versus cold knife. Am J Rhinol Allergy. 2014 Nov-Dec;28(6):517-9. doi: 10.2500/ajra.2014.28.4109. PMID 25514489